CLINICAL TRIAL: NCT02115347
Title: A Phase 1, Non-randomized, Open-label, Single Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Ertugliflozin (MK-8835/PF-04971729) in Subjects With Hepatic Impairment and the Healthy Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics, Safety, and Tolerability of Ertugliflozin (MK-8835/PF-04971729) in Participants With Hepatic Impairment and in Healthy Participants (MK-8835-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8835-014; MK-8835-014 (Other: Merck Study number); B1521024 (Other: Pfizer Study number)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus; Hepatic Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ertugliflozin 15 mg - Moderate Hepatic Impairment (Experimental): Participants receive a single 15 mg oral dose (tablet) of ertugliflozin
  Interventions: Drug: Ertugliflozin 15 mg
- Ertugliflozin 15 mg - Healthy Participants (Other): Participants receive a single 15 mg oral dose (tablet) of ertugliflozin
  Interventions: Drug: Ertugliflozin 15 mg
- Ertugliflozin 15 mg - Mild Hepatic Impairment (Experimental): Participants receive a single 15 mg oral dose (tablet) of ertugliflozin
  Interventions: Drug: Ertugliflozin 15 mg

INTERVENTIONS:
Drug: Ertugliflozin 15 mg — Tablet

SUMMARY:
This is a study to assess the pharmacokinetics and safety of ertugliflozin (MK-8835, PF-04971729) in participants with hepatic impairment versus healthy participants. In Part 1 of the study, participants with moderate hepatic impairment (Child-Pugh score 7-9) and matched healthy participants will be enrolled; depending on results in Part 1, Part 2 may be conducted and will enroll participants with mild hepatic impairment (Child-Pugh score 5-6).

ELIGIBILITY:
Inclusion Criteria:

ALL PARTICIPANTS:

* Body Mass Index (BMI) of 18 to 40 kg/m^2; and a total body weight >50 kg (110 lbs)
* Male or female not of reproductive potential
* If a female of reproductive potential, agrees to remain abstinent from heterosexual activity or agree to use or have their partner use 2 methods of acceptable contraception to prevent pregnancy while the participant is receiving study medication and for 14 days after the last dose of study medication PARTICIPANTS WITH NORMAL HEPATIC FUNCTION
* Healthy with normal hepatic function PARTICIPANTS WITH HEPATIC IMPAIRMENT
* Satisfy the criteria for Child-Pugh classification [moderate (Part 1): Child-Pugh Scores 7-9 points, mild (Part 2): Child-Pugh Scores 5-6 points] within 14 days before administration of study medication
* A diagnosis of hepatic impairment due to primary liver disease and not secondary to other diseases
* Stable hepatic impairment, defined as no clinically-significant change in disease status within the last 30 days
* On a stable dose of medication and/or treatment regimen used to manage hepatic disease for at least 4 weeks prior to study start

Exclusion Criteria:

ALL PARTICIPANTS

* A known hypersensitivity or intolerance to ertugliflozin or any other Sodium-Glucose co-Transporter 2 (SGLT2) inhibitor (i.e., canagliflozin [Invokana], dapagliflozin [Farxiga], empagliflozin, or ipragliflozin)
* Febrile illness within 5 days prior to the first dose of study medication
* Any clinically significant malabsorption condition
* A positive urine drug screen for drugs of abuse or recreational drugs
* Abuse of alcohol or binge drinking and/or any other illicit drug use or dependence within 6 months of study start
* Treatment with an investigational drug within 30 days preceding the first dose of study medication
* Pregnant or breastfeeding females
* Use of herbal supplements within 28 days prior to the first dose of study medication
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing
* History of sensitivity to heparin or heparin-induced thrombocytopenia PARTICIPANTS WITH NORMAL HEPATIC FUNCTION
* Use of prescription drugs (hormonal methods of birth control are allowed), vitamins, and dietary supplements within 7 days prior to the first dose of study medication
* Positive serology for Hepatitis B or C PARTICIPANTS WITH HEPATIC IMPAIRMENT
* Hepatic carcinoma and hepatorenal syndrome or life expectancy less than 1 year
* Undergone portal-caval shunt surgery
* History of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than 1 month prior to study entry
* Signs of significant hepatic encephalopathy
* Severe ascites and/or pleural effusion
* A transplanted kidney, heart or liver
* Received any of the following medications within 7 days prior to the first dose of study medication or during the study: other SGLT2 inhibitors (eg, dapagliflozin, canagliflozin, empagliflozin, and ipragliflozin); any potent drug-metabolizing enzyme-inducing drug, including rifampin, phenytoin, and carbamazepine; probenecid, valproic acid, gemfibrozil

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2015-01-10 (Actual); Study Completion 2015-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck/Pfizer

REFERENCES:
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736
- [Derived] Sahasrabudhe V, Terra SG, Hickman A, Saur D, Raje S, Shi H, Matschke K, Zhou S, Cutler DL. Pharmacokinetics of Single-dose Ertugliflozin in Patients With Hepatic Impairment. Clin Ther. 2018 Oct;40(10):1701-1710. doi: 10.1016/j.clinthera.2018.06.015. Epub 2018 Sep 14. PMID 30224193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Based on a statistical evaluation of the pharmacokinetic (PK) data obtained from participants with moderate hepatic impairment and matched healthy volunteers, and the pre-specified decision criteria, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Groups:
- Ertugliflozin 15 mg (Moderate Hepatic Impairment); Ertugliflozin 15 mg (Normal Hepatic Function): Participants received a single 15 mg oral dose (tablet) of ertugliflozin.
Period: Overall Study
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function) | Ertugliflozin 15 mg - Mild Hepatic Impairment
Started | 8 | 8 | 0
Completed | 8 | 8 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PK concentration population was defined as all participants treated who had at least 1 concentration measurement. Based on evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Full Range); unit: Years] | 55.1 (3.4) [49 to 60] | 55.5 (3.0) [51 to 59] | 55.3 [49 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUClast) for Ertugliflozin
Description: Area under the plasma concentration-time profile from time zero to time of the last quantifiable concentration (AUClast).
Time Frame: Hour 0 (predose), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours
Population: The analysis population was all treated participants who had at least 1 measurement of the AUClast parameter. Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Number analyzed (Participants) | 8 | 8
ng•hr/mL | 1413 (39) | 1618 (14)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Moderate Hepatic Impairment) vs Ertugliflozin 15 mg (Normal Hepatic Function); Test type: Superiority or Other; Ratio (Test/Reference) of Adjusted Means = 87.31, 90% CI 2-sided [68.01 to 112.08] — ANOVA model with hepatic function group as a fixed effect, ratios (and 90% confidence intervals [CIs]) were expressed as percentages, Moderate Hepatic Impairment (Test), Normal Hepatic Function (Reference)

2. Primary Outcome: AUC From Hour 0 to Infinity (AUCinf) for Ertugliflozin
Description: Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf).
Time Frame: Hour 0 (predose), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours
Population: The analysis population was all treated participants who had at least 1 measurement of the AUCinf parameter. Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Number analyzed (Participants) | 8 | 8
ng•hr/mL | 1430 (39) | 1636 (14)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Moderate Hepatic Impairment) vs Ertugliflozin 15 mg (Normal Hepatic Function); Test type: Superiority or Other; Ratio (Test/Reference) of Adjusted Means = 87.43, 90% CI 2-sided [68.11 to 112.22] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUClast for Fraction of Ertugliflozin Unbound in Plasma (AUClast,u)
Description: Area under the plasma concentration-time profile from time zero to time of the last quantifiable concentration (Clast) for unbound drug (ertugliflozin only).
Time Frame: Hour 0 (predose), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours
Population: The analysis population was all treated participants who had at least 1 measurement of the AUClast,u parameter. Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Number analyzed (Participants) | 8 | 8
ng•hr/mL | 52.47 (44) | 54.77 (15)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Moderate Hepatic Impairment) vs Ertugliflozin 15 mg (Normal Hepatic Function); Test type: Superiority or Other; Ratio (Test/Reference) of Adjusted Means = 95.81, 90% CI 2-sided [72.40 to 126.79] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: AUCinf for Fraction of Ertugliflozin Unbound in Plasma (AUCinf,u)
Description: Area under the plasma concentration-time profile from time zero extrapolated to infinite time for unbound drug (ertugliflozin only) (AUCinf, u).
Time Frame: Hour 0 (predose), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours
Population: The analysis population was all treated participants who had at least 1 measurement of the AUCinf,u parameter. Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Number analyzed (Participants) | 8 | 8
ng•hr/mL | 53.14 (44) | 55.40 (16)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Moderate Hepatic Impairment) vs Ertugliflozin 15 mg (Normal Hepatic Function); Test type: Superiority or Other; Ratio (Test/Reference) of Adjusted Means = 95.92, 90% CI 2-sided [72.46 to 126.97] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Ertugliflozin
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given.
Time Frame: Hour 0 (predose), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours
Population: The analysis population was all treated participants who had at least 1 measurement of the Cmax parameter. Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Number analyzed (Participants) | 8 | 8
ng/mL | 251.1 (27) | 319.0 (11)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Moderate Hepatic Impairment) vs Ertugliflozin 15 mg (Normal Hepatic Function); Test type: Superiority or Other; Ratio (Test/Reference) of Adjusted Means = 78.70, 90% CI 2-sided [65.74 to 94.23] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Cmax for Fraction of Ertugliflozin Unbound in Plasma (Cmax,u)
Description: Maximum plasma concentration for unbound drug (ertugliflozin only).
Time Frame: Hour 0 (predose), and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, and 96 hours
Population: The analysis population was all treated participants who had at least 1 measurement of the Cmax,u parameter. Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Number analyzed (Participants) | 8 | 8
ng/mL | 9.336 (30) | 10.79 (15)
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg (Moderate Hepatic Impairment) vs Ertugliflozin 15 mg (Normal Hepatic Function); Test type: Superiority or Other; Ratio (Test/Reference) of Adjusted Means = 86.52, 90% CI 2-sided [70.49 to 106.20] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 19 days
Population: The analysis population was defined as all treated participants. Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Measure: Number; unit: Participants
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Number analyzed (Participants) | 8 | 8
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to Day 19
Description: Based on a statistical evaluation of the PK data from participants with moderate hepatic impairment and matched healthy volunteers, Part 2 of the study was not conducted and participants with mild hepatic impairment were not enrolled.
Arm/Group | Ertugliflozin 15 mg (Moderate Hepatic Impairment) | Ertugliflozin 15 mg (Normal Hepatic Function)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 15 mg (Moderate Hepatic Impairment) (N=8) | Ertugliflozin 15 mg (Normal Hepatic Function) (N=8)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to the sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.